CLINICAL TRIAL: NCT07119918
Title: PCSK9 Inhibitor for Intracranial Atherosclerotic Symptomatic Stenosis (PICASSO): A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: PCSK9 Inhibitor for Intracranial Atherosclerotic Symptomatic Stenosis
Acronym: PICASSO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Vice President of Sun Yat-sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PICASSO
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Symptomatic Intracranial Atherosclerotic Stenosis
Keywords: symptomatic intracranial atherosclerotic stenosis; Recaticimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recaticimab group (Experimental)
  Interventions: Drug: Recaticimab
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recaticimab — Recaticimab 300mg subcutaneous Q8W for 1 year.
  Arms: Recaticimab group
Drug: Placebo — Matched placebo subcutaneous Q8W for 1 year.
  Arms: Placebo group

SUMMARY:
An investigator-initiated, prospective, multicenter, randomized, double-blind, placebo-controlled trial comparing the 1-year incidence of stroke in patients with AIS or TIA within 7 days who are treated with either placebo or Recaticimab.

DETAILED DESCRIPTION:
This is an investigator-initiated, prospective, multicenter, randomized, double-blind, placebo-controlled trial to determine the efficacy of Recaticimab (PCSK9 inhibitor) administered within 7 days of symptom onset in patients with symptomatic intracranial atherosclerotic stenosis (sICAS) in reducing incident stroke within 1 year.

Study intervention: (1) Participants in the intervention group will receive Recaticimab 300mg subcutaneous Q8W for 1 year. (2) Participants in the control group will receive matched placebo subcutaneous Q8W for 1 year. All participants will receive best medical management (BMM), including intensive statins treatment and dual antiplatelet therapy.

A total of 5276 participants are anticipated to be recruited for this study. Eligible participants will be 1:1 randomly assigned to receive Recaticimab or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥30 years and ≤80 years.

Patients aged between 30 to 49 are required to meet at least one of the following criteria:

1. Insulin dependent diabetes for at least 15 years.
2. At least 2 of the following atherosclerotic risk factors: hypertension (BP > 140/90 or on antihypertensive therapy); dyslipidemia (LDL > 130 mg /dL or HDL < 40 mg/dL or fasting triglycerides > 150 mg/dL or on lipid lowering therapy); smoking; non-insulin dependent diabetes or insulin dependent diabetes of less than 15 years duration; family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery in parent or sibling who was < 55 years of age for men or < 65 for women at the time of the event.
3. History of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease.
4. Any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic.
5. Aortic arch atheroma documented by non-invasive vascular imaging or catheter angiography vi. any aortic aneurysm documented by non-invasive vascular imaging or catheter angiography that is considered atherosclerotic.

2. Diagnosed with acute ischemic stroke or moderate-to-high risk transient ischemic attack (ABCD2 score ≥4).

3. CTA or DSA confirmed intracranial atherosclerotic stenosis >50%, which was responsible for the incident.

4. The time from symptom onset to initiation of study treatment is within 7 days.

5. Signed informed consent.

Exclusion Criteria:

1. Baseline NIHSS ≥26.
2. Suspected cardiogenic ischemic cerebrovascular diseases (e.g., combined with atrial fibrillation, heart valve prosthesis, atrial myxoma, endocarditis, etc.).
3. Source of symptoms is possible related to ipsilateral carotid disease.
4. Other ischemic cerebrovascular diseases with specific causes (e.g., aortic dissection, vasculitis, vascular malformation, etc.).
5. Non-cerebral vascular disease (e.g., intracranial tumors, multiple sclerosis).
6. Hemorrhagic stroke or hemorrhagic transformation of cerebral infarction before randomization.
7. Pre-existing contraindications of using PCSK9 inhibitors.
8. Use of any PCSK9 inhibitors within the past 3 months.
9. Pregnant or childbearing-age women who have no effective contraceptives or positive pregnancy test records.
10. Patients who are participating in other trials.
11. Hepatic or renal dysfunction, defined as AST and/or ALT >3ULN，eGFR<30mL/min, or Crea >220μmol/L (2.5mg/dL).
12. Uncontrolled hypertension defined as systolic blood pressure (BP) >220mmHg or diastolic BP >120mmHg.
13. Life expectancy is less than 1 year due to severe non-cardiovascular disease.
14. Angioplasty or stenting procedure is planned before randomization.
15. Unable to finish the follow-up visit due to geographical factor or other reasons (e.g., dementia, alcoholism, substance abuse, severe mental disease, etc.)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5276 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Any new stroke | 1 year (±2) weeks
  Any new ischemic or hemorrhagic stroke within 1 year

SECONDARY OUTCOMES:
Composite cardiovascular events | 1 year (±2) weeks
  Composite cardiovascular events (non-fatal stroke, myocardial infarction, and death from cardiovascular causes) within 1 year.
Ischemic stroke | 1 year (±2) weeks
  Any new ischemic stroke within 1 year.
Hemorrhagic stroke | 1 year (±2) weeks
  Any new hemorrhagic stroke within 1 year.
Non-fatal stroke | 1 year (±2) weeks
  Any non-fatal stroke within 1 year.
Myocardial infarction | 1 year (±2) weeks
  Any myocardial infarction within 1 year.
Death from cardiovascular causes | 1 year (±2) weeks
  Any death from cardiovascular causes within 1 year.
Quality of life (EQ-5D-5L) | 1 year (±2) weeks
  1-year quality of life measured by EQ-5D-5L.
NIHSS scores | 7(±1) days or discharge
  NIHSS scores at 7 days or discharge.
Modified Rankin Scale score at 90 days | 90 (±14) days
  The shift analysis of the 90-day mRS at 90 days.
Modified Rankin Scale score at 1 year | 1 year (±2) weeks
  The shift analysis of the 90-day mRS at 1 year.
Safety outcome: intracranial hemorrhage | 1 year (±2) weeks
  Symptomatic intracranial hemorrhage within 1 year.
Safety outcome: Death | 1 year (±2) weeks
  Death within 1 year.
Safety outcome: Serious Adverse Event (SAE) | 1 year (±2) weeks
  Any SAE within 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from Principal Investigators (Prof. Yamei Tang) upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the trial completion.
Access Criteria: The IPD will be available from Principal Investigators (Prof. Yamei Tang) upon reasonable request.